CLINICAL TRIAL: NCT05092386
Title: An Open-label Combined Randomized Double-blind, Positive Control Clinical Trial in Subjects Aged 2 Months (Minimum 6 Weeks) and Above to Preliminary Evaluate the Safety and Immunogenicity of a 13-valent Pneumococcal Polysaccharide Conjugate Vaccine
Brief Title: Safety and Immunogenicity Study of a 13-valent Pneumococcal Polysaccharide Conjugate Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-PCV-1001
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Open label design will be adopted for children and adolescents aged 6-17 years and infants aged 3 months, and randomized, blind and positive control design was adopted for other populations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Experimental Group of One Dose (Experimental): 110 Participants (including 20 subjects aged 18~49 years, 20 subjects aged 6~17 years , 30 subjects aged2-5 years) will receive one dose of experimental vaccine
  Interventions: Biological: Investigational 13-valent Pneumococcal Polysaccharide Conjugate Vaccine
- Experimental Group of Two Doses (Experimental): 30 Participants aged 12~23 months will receive two doses of experimental vaccine on the schedule of month 0,2.
  Interventions: Biological: Investigational 13-valent Pneumococcal Polysaccharide Conjugate Vaccine
- Experimental Group of Three Doses (Experimental): 30 Participants aged 7~11 months will receive two doses of experimental vaccine on the primary immunization schedule of month 0,2 and one dose of booster immunization during the participants aged 12~15 months .
  Interventions: Biological: Investigational 13-valent Pneumococcal Polysaccharide Conjugate Vaccine
- Experimental Group of Four Doses (Experimental): 30 Participants aged 3 months will receive three doses of experimental vaccine on the primary immunization schedule of month 0,1,2 and one dose of booster immunization during the participants aged 12~15 months ; 30 Participants aged 2 months will receive three doses of experimental vaccine on the primary immunization schedule of month 0,2,4 and one dose of booster immunization during the participants aged 12~15 months
  Interventions: Biological: Investigational 13-valent Pneumococcal Polysaccharide Conjugate Vaccine
- Control Group of One Dose With WALVAX PCV13 (Active Comparator): 30 Participants aged 2-5 years will receive one dose of control vaccine (WALVAX PCV13)
  Interventions: Biological: Control 13-valent Pneumococcal Polysaccharide Conjugate Vaccine ( WALVAX PCV13)
- Control Group of Two Doses With WALVAX PCV13 (Active Comparator): 30 Participants aged 12~23 months will receive two doses of control vaccine(WALVAX PCV13) on the schedule of month 0,2.
  Interventions: Biological: Control 13-valent Pneumococcal Polysaccharide Conjugate Vaccine ( WALVAX PCV13)
- Control Group of Three Doses With WALVAX PCV13 (Active Comparator): 30 Participants aged 7~11 months will receive two doses of control vaccine(WALVAX PCV13) on the primary immunization schedule of month 0,2 and one dose of booster immunization during the participants aged 12~15 months .
  Interventions: Biological: Control 13-valent Pneumococcal Polysaccharide Conjugate Vaccine ( WALVAX PCV13)
- Control Group of Three Doses With Pfizer PCV13 (Active Comparator): 30 Participants aged 2 months will receive three doses of control vaccine(Pfizer PCV13 on the primary immunization schedule of month 0,2,4 and one dose of booster immunization during the participants aged 12~15 months
  Interventions: Biological: Control 13-valent Pneumococcal Polysaccharide Conjugate Vaccine ( Pfizer PCV13)

INTERVENTIONS:
Biological: Investigational 13-valent Pneumococcal Polysaccharide Conjugate Vaccine — The investigational vaccine was manufactured by Sinovac Research & Development Co., Ltd. each for purified 13 serotypes of pneumococcal polysaccharide and diphtheria CRM197 in 0·5 mL of aluminum phosphate ,sodium chloride,polysorbate 80 and succinic acid per injection.
  Arms: Experimental Group of Four Doses; Experimental Group of One Dose; Experimental Group of Three Doses; Experimental Group of Two Doses
Biological: Control 13-valent Pneumococcal Polysaccharide Conjugate Vaccine ( WALVAX PCV13) — The control vaccine was manufactured by WALVAX Biotechnology Co., Ltd. each for purified 13 serotypes of pneumococcal polysaccharide and tetanus toxoid vector (TT) in 0·5 mL of aluminum phosphate ,disodium hydrogen phosphate and sodium dihydrogen phosphate per injection.
  Arms: Control Group of One Dose With WALVAX PCV13; Control Group of Three Doses With WALVAX PCV13; Control Group of Two Doses With WALVAX PCV13
Biological: Control 13-valent Pneumococcal Polysaccharide Conjugate Vaccine ( Pfizer PCV13) — The control vaccine was manufactured by Pfizer. each for purified 13 serotypes of pneumococcal polysaccharide and tetanus toxoid vector (TT) in 0·5 mL of aluminum phosphate ,sodium chloride ,succinic acid ,polysorbate 80 and water for injection per injection.
  Arms: Control Group of Three Doses With Pfizer PCV13

SUMMARY:
This study is an open-label combined randomized double-blind, positive control phase Ⅰ clinical trial of the a 13-valent Pneumococcal Polysaccharide Conjugate Vaccine manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to preliminary evaluate the safety and immunogenicity of the study vaccine

DETAILED DESCRIPTION:
This study is an open-label combined randomized double-blind, positive control phase Ⅰ clinical trial in subjects aged 2 months (minimum 6 weeks) and above. The experimental vaccine was manufactured by Sinovac Research & Development Co., Ltd. .And one of the positive control vaccine was manufactured by WALVAX Biotechnology Co., Ltd( WALVAX PCV13) ,the other manufactured by Pfizer(Pfizer PCV13).A total of 310 subjects including 20 adults aged 18-49 years,20 adolescents and children aged 6~7 years ,60 children aged 2-5 years,60 infants aged 12~23 months,60 infants aged 7 ~11 months,60 infants aged 2 months (minimum 6 weeks), and 30 infants aged 3 months will be enrolled.Subjects will be assigned to receive one dose , two doses ,three doses or four doses of experimental vaccine or different positive control vaccines . Subjects aged 18-49 years will receive one dose of experimental vaccine.Subjects aged 6~17 years will receive one dose of experimental vaccine.Subjects aged 2~5 years will be randomly divided into two groups in a ratio of 1:1,and each group will receive one dose of experimental vaccine or control vaccine(WALVAX PCV13）.Subjects aged 7 ~ 11 months and subjects aged 12 ~23 months will be randomly divided into two groups in a 1:1 ratio,the subjects aged 12 ~ 23 months will receive two doses of experimental vaccine or control vaccine on the schedule of month 0,2 .Subjects aged 7 ~11 months will receive 3 doses of experimental vaccine or control vaccine (WALVAX PCV13）on the immunization schedule of month 0,2,4.Subjects aged 3 months will receive 4 doses of experimental vaccine.Subjects aged 2 months will be randomly divided into 2 groups in a 1:1 ratio and each group will receive 4 doses of experimental vaccine or control vaccine (Pfizer PCV13).

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 2 months (minimum 6 weeks), healthy infants aged 3 months, healthy infants aged 7 ~ 11 months, healthy infants aged 12~ 23 months, healthy children aged 2~ 5 years, healthy adolescent and children aged 6~ 17 years, healthy adults aged 18~ 49 years；
* Proven legal identification and vaccination certificate (vaccination certificate is required for those aged 5 and below)；
* The subject and/or guardian can understand and voluntarily sign the informed consent form.

Exclusion Criteria:

* Have received pneumococcal polysaccharide vaccine or pneumococcal polysaccharide conjugate vaccine;
* Have Bacterial pneumonia or invasive pneumococcal infectious disease (IPD) caused by pneumococcus confirmed by sputum culture;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* History of thyroidectomy, absence of spleen, functional absence of spleen, and absence of spleen or splenectomy due to any circumstance;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute diseases or acute exacerbation of chronic diseases in the past 7 days;
* Axillary temperature >37.0°C;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 6 Weeks to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 310 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-05-26 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Safety index-incidence of adverse reactions | Day 0-30 after each dose of experimental vaccine
  Incidence of adverse reactions 0 to 30 days after each dose of experimental vaccine

SECONDARY OUTCOMES:
Safety index-incidence of adverse reactions | Day 0-7 after each dose of experimental vaccine
  Incidence of adverse reactions 0 to 7 days after each dose of experimental vaccine
Safety index-incidence of abnormal indicators | Day 3 after vaccination after each dose of experimental vaccine
  Incidence of abnormal indicators of Blood routine, blood biochemistry and urine routine 3 days after vaccination in subjects aged 2 years and older
Safety index-Incidence of serious adverse events during the safety observation period | 1 month after vaccination ,6 months after primary immunization or 1 month after booster immunization
  Incidence of serious adverse events during the safety observation period, including 1 month after vaccination in subject aged 6 years and older, and 6 months after primary immunization and 1 month after booster immunization in subject aged 2 months (minimum 6 weeks) to 5 years(if any)
Immunogenicity index-Geometric mean concentrations (GMC) and GMI of specific IgG for each serotype | Day 30 after vaccination
  Geometric mean concentrations (GMC) and GMI of specific IgG for each serotype at 30 days after vaccination in subjects of all age groups
Immunogenicity index-Geometric mean titers (GMT) and GMI of serotype specific opsonophagocytic antibody OPA for each serotype | Day 30 after vaccination
  Geometric mean titers (GMT) and GMI of serotype specific opsonophagocytic antibody OPA for each serotype at 30 days after vaccination in subjects of all age groups
Immunogenicity index-Seropositive rates，GMCs and GMI of serum specific antibody | Day 30 after vaccination
  Seropositive rates of IgG concentration ≥0.35μg/mL, ≥1.0μg/mL, geometric mean concentration (GMCs) and GMI of serum specific antibody at 30 days after primary immunization in subjects of all age groups
Immunogenicity index-Proportion of OPA ≥1:8 of each serum and geometric mean titer (GMT) | Day 30 after vaccination
  Proportion of OPA ≥1:8 of each serum and geometric mean titer (GMT)in subjects of all age groups at 30 days after primary immunization
Immunogenicity index-Seropositive rates of IgG concentration ≥0.35μg/mL, ≥1.0μg/mL, geometric mean concentration (GMC) | Day 30 before and after booster immunization
  Seropositive rates of IgG concentration ≥0.35μg/mL, ≥1.0μg/mL, geometric mean concentration (GMC) in subjects aged 2 months (Minimum 6 weeks), 3 months and 7 ~ 11 months at 30 days before and after booster immunization
Immunogenicity index-Proportion of OPA ≥1:8 for each serotype and geometric mean titer (GMT) | Day 30 before and after booster immunization
  Proportion of OPA ≥1:8 for each serotype and geometric mean titer (GMT) in subjects aged 2 months (Minimum 6 weeks), 3 months, and 7~ 11 months at 30 days before and after booster immunization

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Master, Principal Investigator — Henan Provincial Center for Disease Prevention and Control
Locations (1):
- Henan Center for Diseases Control and Prevention, Zhengzhou, Henan, China